CLINICAL TRIAL: NCT00647153
Title: Pre-Surgical Detection of Colorectal Carcinomas Using 123Iodine-Labeled cT84.66 Diabody Antibody Fragments to Carcinoembryonic Antigen (CEA)
Brief Title: Immunoscintigraphy Using Radiolabeled Monoclonal Antibody in Finding Tumor Cells in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04085; P30CA033572 (NIH); CHNMC-04085; CDR0000590136 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-03-28; First posted 2008-03-31 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation: iodine I 123 anti-CEA recombinant diabody T84.66 (Experimental)
  Interventions: Other: pharmacological study; Procedure: single photon emission computed tomography; Radiation: iodine I 123 anti-CEA recombinant diabody T84.66

INTERVENTIONS:
Other: pharmacological study — Pre-infusion and 30 min., 1h,2h, and 3-4h post start of infusion. Day 1 and 2 post infusion.
Procedure: single photon emission computed tomography — One day post infusion
Radiation: iodine I 123 anti-CEA recombinant diabody T84.66 — 10mCi/mg

SUMMARY:
RATIONALE: Diagnostic procedures, such as immunoscintigraphy, using a radiolabeled monoclonal antibody may help find and diagnose colorectal cancer.

PURPOSE: This clinical trial is studying how well immunoscintigraphy using a radiolabeled monoclonal antibody works in finding tumor cells in patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the ability of iodine I 123 anti-CEA recombinant diabody T84.66 to localize to colorectal cancer, as determined by quantitative radioimmunoscintigraphy in patients with colorectal cancer.

Secondary

* To evaluate the clinical pharmacokinetics of iodine I 123 anti-CEA recombinant diabody T84.66 clearance in these patients.
* To characterize the frequency and titer of the human anti-chimeric response to iodine I 123 anti-CEA recombinant diabody T84.66 in these patients.
* To determine the safety of iodine I 123 anti-CEA recombinant diabody T84.66 in these patients.

OUTLINE: Patients receive an infusion of iodine I 123 anti-CEA recombinant diabody T84.66. Patients undergo planar imaging every 5 minutes during the radiolabeled antibody infusion and then at 3-6 hrs, 12-24 hours, and, if indicated, 30-48 hours after the radiolabeled antibody infusion. Planar spot images of the head, chest, abdomen, and pelvis and whole body images (anterior and posterior) are taken. Patients also undergo SPECT scan of the abdomen and pelvis at 12 and 24 hours after the radiolabeled antibody infusion.

Blood samples are collected for pharmacokinetic analysis immediately after the radiolabeled antibody infusion and then at 15 minutes, 30 minutes, 1 hour, 2 hours, and 4 hours after the radiolabeled antibody infusion.

Patients are followed periodically for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Stage I-IV disease

PATIENT CHARACTERISTICS:

* Serum creatinine < 2.0 mg/dL
* Total bilirubin < 2.0 mg/dL
* Hemoglobin > 9.0 g/dL
* cT84.66 antibody negative (if previously treated with mouse or chimeric immunoglobulins)
* Not pregnant
* No condition that, in the opinion of the investigator, would preclude study compliance
* No known allergy to iodine
* No known history of HIV, hepatitis B, or hepatitis C

PRIOR CONCURRENT THERAPY:

* No concurrent steroids

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Tumor targeting properties of iodine I 123 anti-CEA recombinant diabody T84.66 | Day 2 post infusion

SECONDARY OUTCOMES:
Clinical pharmacokinetics of iodine I 123 anti-CEA recombinant diabody T84.66 | Day 2 post infusion
Immunogenicity properties of iodine I 123 anti-CEA recombinant diabody T84.66 | 6 months post infusion
Safety of iodine I 123 anti-CEA recombinant diabody T84.66 | 6 months post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y. Wong, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States